CLINICAL TRIAL: NCT00830895
Title: A Phase II Study to Evaluate the Efficacy of RAD001 in Metastatic Non-clear Cell Renal Cell Carcinoma
Brief Title: RAD001 for Non-clear Cell Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-RENAL-0901
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Non-clear cell; RAD001; Metastatic, non-clear cell, renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): RAD001 10mg/day
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 10mg/day

SUMMARY:
To assess the efficacy and safety of RAD001 (everolimus) in non-clear cell renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-clear cell renal cell carcinoma (papillary, chromophobe, collecting duct, oncocytic subtype, sarcomatoid mainly)
2. Subjects with metastatic legion
3. Subjects aged 18 years or older
4. Subjects whose ECOG performance status is 0 or 1
5. Subjects who have laboratory value below; Hematology

   * Neutrophil >= 1.5 x 109/L
   * Platelet >= 75 x 109/L
   * Hemoglobin >= 9 g/dL Liver function tests
   * Total bilirubin ≤ 1.5 xULN
   * AST, ALT ≤ 2.5 xULN
   * Alkaline phosphatase ≤ 2.5 xULN Renal function tests
   * Creatinine clearance >= 30 mL/min
6. Subjects who understand and provide a written informed consent

Exclusion Criteria:

1. Subjects who have been administered an mTOR inhibitor
2. Pregnant or nursing women, and women of childbearing potential must use appropriate contraception for the study period and the result of their pregnancy test performed within 14 days before enrollment must be negative
3. Subjects who participated in a clinical study using the study medication within 30 days before randomization
4. Subjects with clinically uncontrolled central nervous system (CNS) metastasis
5. Subjects with life expectancy of less than 3 months
6. Subjects with interstitial pulmonary disease
7. Subjects whose QTc interval is prolonged (QTc > 450 msec for male or > 470 msec for female)
8. Other serious diseases or medical conditions Heart disease unstable despite treatment History of myocardial infarction within six months before the study History of serious neurological or psychological disorder including dementia or seizure Active peptic ulcer which cannot be controlled by a drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 months, 4 months, 6 months
  It is the time from treatment initiation until disease progression.

SECONDARY OUTCOMES:
Response rate | 2 months, 4 months, 6 months
  It is the percentage of patients whose cancer shrinks or disappears after treatment.
Disease-control rate | 2 months, 4 months, 6 months
  It is the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention.
Overall survival | 2 months, 4 months, 6 months
  The length of time from either the date of diagnosis or the start of treatment for a disease that patients diagnosed with the disease are still alive.
Metabolic response rate by FDG-PET | 2 months, 4 months, 6 months
  It is assesed target lesions and non- target lesions by FDG-PET.
Safety | monthly

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Koh Y, Lim HY, Ahn JH, Lee JL, Rha SY, Kim YJ, Kim TM, Lee SH. Phase II trial of everolimus for the treatment of nonclear-cell renal cell carcinoma. Ann Oncol. 2013 Apr;24(4):1026-31. doi: 10.1093/annonc/mds582. Epub 2012 Nov 23. PMID 23180114